CLINICAL TRIAL: NCT06468345
Title: The Effect of Acupressure Applied After Bariatric Surgery on Gastrointestinal Functions, Pain and Anxiety
Brief Title: Acupressure Application in Obesity Surgery 2345
Acronym: DB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Duygu Balaban, Chief investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DBalaban
Record Dates: First submitted 2024-05-22; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acupressure; Bariatric Surgery; Spleen Meridian; Pregnancy Meridian; Stomach Meridian
MeSH Terms: interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure Group (Experimental): Acupressure application to CV12, ST25, SP6, LI4 and HT7 areas
  Interventions: Behavioral: acupressure
- Control Group (No Intervention): No action was taken.
- Placebo Group (Sham Comparator): Massage application to feet, hands and abdomen areas that are not acupressure areas
  Interventions: Behavioral: Area different from acupressure area

INTERVENTIONS:
Behavioral: acupressure — Application was made to CV12, ST25, SP6, HT7 and LI4 acupressure areas.
  Arms: Acupressure Group
Behavioral: Area different from acupressure area — Massage application to non-acupressure hand, foot and abdominal areas
  Arms: Placebo Group

SUMMARY:
This research was conducted to determine the effect of acupressure applied to patients after bariatric surgery on gastrointestinal distress, pain and anxiety. The data of the study was collected at Aktif Private Kocaeli Hospital General Surgery Clinic between January 2022 and February 2023. The study was conducted with 90 (30 control, 30 intervention and 30 placebo) patients who underwent bariatric surgery. As a result of the research, application to ST25 and CV12 acupressure areas after bariatric surgery increased gas and stool output. It reduced abdominal distension. This enabled patients to start oral intake early. Application to the SP6 area reduced abdominal pain. Acupressure applied to the LI4 area was not effective in reducing nausea and vomiting. Massage to the HT7 acupressure area alone was not sufficient to relieve anxiety.

DETAILED DESCRIPTION:
This research was conducted to determine the intensity of acupressure treatment for gastrointestinal problems, pain and anxiety after bariatric surgery. The research was conducted using a placebo group, randomized controlled, detailed research model. The data of the study was collected at Aktif Private Kocaeli Hospital General Surgery Clinic between January 2022 and February 2023. The study was conducted with 90 (30 control, 30 intervention and 30 placebo) patients who underwent bariatric surgery. The data were brought together with the patient identification formula, postoperative gastrointestinal functions information formula, abdominal distension formula, visual analog scale, state-trait anxiety inventory scale, visual comparison operation, and patient happiness formula. The data were analyzed with the SPSS for Windows 22 package program. Records of numbers, percentages, minimum and maximum values, averages and standard deviations in the analysis of data. Mann Whitney U analysis, LSD, Dunnet C, Kruskall Wallis, Will coxon analyzes and t test records. The results were interpreted at the p< 0.05 significance level. Gastrointestinal capacity and recovery time, stool and gas output rates, difference in distension and abdominal pain score amounts, oral intake amounts and retching difference of the patients in acupressure, control and placebo distribution at the 6th, 12th, 24th and 48th months of the surgery were investigated. Children's movements and vomiting were evaluated with visual comparison performance. Anxiety was measured with the State-Trait Anxiety Inventory Scale at the ages of 6, 12, 24 and 48 after treatment. He recorded the Patient Satisfaction Form to obtain the patients' satisfaction after acupressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Bariatric Surgery
* Conscious patients between the ages of 18-65
* Patients who can communicate
* Patients without hearing-speech problems
* Patients without any psychiatric disorder
* Patients willing to cooperate
* Patients who have never had acupressure before
* Patients who do not have conditions such as hematoma, wound or fracture in the areas where acupressure will be applied

Exclusion Criteria:

* Patients who withdraw from the study at any stage of the study
* Patients admitted to the intensive care unit in the early postoperative period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain after obesity surgery in the intervention, placebo and control groups with the Visual Analog pain scale | Pain was assessed at 24 hours postoperatively.
  On the Visual Analog pain scale, a score of 0 means no pain and 10 means unbearable pain.

SECONDARY OUTCOMES:
Evaluating the distension of patients after obesity surgery with the Abdominal Distension Form | Distention of the patients was measured at the 24th postoperative hour.
  The Abdominal Distension Form ranges from 0 to no distension and 10 to severe distension.

OTHER OUTCOMES:
Measuring the gastrointestinal functions of patients after obesity surgery with the Gastrointestinal Functions Information Form | Gastrointestinal functions of the patients were measured at 6, 12, 24 and 48 hours after surgery.
  The Gastrointestinal Functions Information Form includes a total of 6 questions about the patients' stool output, gas output, oral intake amount, nausea, vomiting and retching. Patients have two ways of answering: yes or no.
Measuring nausea and vomiting in patients after obesity surgery with the Visual Comparison Scale. | Measurements were taken at 6, 12, 24 and 48 hours after surgery.
  In the Visual Comparison Scale, the lowest value of the patients' nausea and vomiting was used as 0 mm, and the highest value was 100 mm.
Measuring the anxiety of patients after bariatric surgery with the State-Trait Anxiety Inventory. | The patients' anxiety was measured at the 24th hour after surgery.
  There are two forms in the State-Trait Anxiety Inventory questionnaire. The first form consists of 20 questions measuring the state anxiety of the patients, and the second form contains 20 questions measuring the trait anxiety of the patients. The lowest score in these questions is 1 and the highest score is 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Üniversitesi, Erzurum, Turkey (Türkiye)